CLINICAL TRIAL: NCT04381611
Title: INTEGRAL Study: A Longitudinal Study of Surgeries and Lasers in Glaucoma: Long-term Results and Success Predictors Analysed From a Large-scale Retrospective and Prospective Glaucoma Register
Status: Enrolling by invitation | Type: Observational
Sponsor: Dr. Kaweh Mansouri (Other)
Responsible Party: Sponsor-Investigator, Dr. Kaweh Mansouri, Professor UC Denver, Swiss Vision Network
Organization: Swiss Vision Network (Other)
Other Study IDs: INTEGRAL
Record Dates: First submitted 2020-04-30; First posted 2020-05-11 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Glaucoma Open-Angle; Glaucoma Eye; Glaucoma; Drugs; Glaucoma, Angle-Closure; Glaucoma Secondary; Glaucoma, Neovascular; Glaucoma Congenital; Surgery; Glaucoma, Pigmentary; Glaucoma Capsulare
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma; Glaucoma, Angle-Closure; Glaucoma, Neovascular; Hydrophthalmos; Exfoliation Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (10):
- Primary Glaucoma
- Glaucoma Surgery
- Glaucoma Laser
- Glaucoma Surgery Combined
- Glaucoma treatment
- Glaucoma imaging
- Glaucoma co-morbidity
- Glaucoma untreated
- Glaucoma Suspect
- Secondary Glaucoma

SUMMARY:
The study is an observational analysis of patients' medical data recorded in a large-scale register, both retrospective (for patients operated and data recorded before 2018) and prospective (for data collected after 2018) in nature.Patients' medical data contained in the register will be analysed to determine the efficacy of the treatments they received during their follow-up at the investigation centre.

DETAILED DESCRIPTION:
This study involves the creation and analysis of a large-scale register including all patients suffering from glaucoma, currently and previously followed-up and treated at a single tertiary centre in Lausanne, Switzerland. The design of the study is longitudinal, observational and comparative. Patients are recruited retrospectively if they attended the research centre before September 2018, and prospectively if they attend the centre from this month onwards. Their inclusion does not affect their care, treatment choice or follow-up. All data of recruited patients is be kept in their medical notes until a specific analysis is launched. Data is then exported from their medical notes into a coded database for analysis. At the end of each analysis session (defined as the publication of the related article), all exported data is fully anonymised.

Data analysis will aim to assess the long-term efficacy, safety profile, and factors predictive of success/failure of treatments performed.

To ensure the quality of all included data, health-related information will be extracted directly from the medical notes and coded into the register by a Clinical Research Associate. Conformity of the process and recorded data will be confirmed by regular internal auditing. For quality assurance the Ethics Committee may visit the research sites. Direct access to the source data and all project related files and documents must be granted on such occasions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of glaucoma (open-angle, closed-angle, primary or secondary) or ocular hypertension (IOP > 24 mmHg, medicated or not)
* Patients who received treatment (medical, laser or surgical) at the Glaucoma Centre, Montchoisi Clinic
* Able and willing to provide informed written or verbal consent

Exclusion Criteria:

* Patient who are unable to understand the implications of their inclusion in the study or who are unable or unwilling to give informed consent

Ages: 1 Year to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Any patient suffering or suspected of glaucoma and treated at Montchoisi Clinic
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2019-01-15 (Actual); Primary Completion 2030-01-15 (Estimated); Study Completion 2030-01-15 (Estimated)

PRIMARY OUTCOMES:
Number of patients with IOP reduction mmHg | 12 month
  Final Intra Ocular Pressure <20% compared to baseline
Patients with quantitative OCT variations ( RNFL, μm) | 12 month
  Variation of RNFL before and after treatment ( laser, surgery, drug..)
Number of patients with quantitative VF variation ( MD, dB) | 12 month
  Visual Field MD variation before and after treatment ( laser, surgery, drug..)
Number of patients with quantitative VF variation (LV, dB) | 12 months
  Visual Field MD variation before and after treatment ( laser, surgery, drug..)

SECONDARY OUTCOMES:
Number of operations received by a patients | 12 month
  Number of operations undertaken by each patient
Number of patients undergoing a specific ocular surgical or laser procedure | 12 month
  Number of patients undertaking different types of ocular procedures ( deep sclerectomy, cataract, LPI, SLT,...)
Number of lowering IOP drugs ( molecules) taken by each patient | 12 month
  Number of molecules used by each patient (e.g Cosopt: 2 molecules, Xalatan: 1...)
Anterior segment OCT variations: ACA (°), SSA (°) | 12 month
  variations of these measurements before and after procedure ( surgery or laser)
Anterior segment OCT variations: AOD (mm) | 12 month
  variations of these measurements before and after procedure ( surgery or laser)
Anterior segment OCT variations: TISA (mm2) | 12 month
  variations of these measurements before and after procedure ( surgery or laser)

CONTACTS AND LOCATIONS:
Locations (1):
- SwissVisio Montchoisi, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Meduri E, Gillmann K, Bravetti GE, Niegowski LJ, Mermoud A, Weinreb RN, Mansouri K. Iridocorneal Angle Assessment After Laser Iridotomy With Swept-source Optical Coherence Tomography. J Glaucoma. 2020 Nov;29(11):1030-1035. doi: 10.1097/IJG.0000000000001654. PMID 32890108